CLINICAL TRIAL: NCT03537625
Title: Effects of Green Tea and Fermented Green Tea Extract on Obese Adults: a Randomized Double-blind, Placebo-controlled Study Focused on Change of Gut Microbiota and Inflammatory Markers
Brief Title: Effects of Green Tea on Body Weight Reduction and Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNUBH-GT
Record Dates: First submitted 2018-04-16; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Green tea (Experimental): Green tea extract 2 gram per day
  Interventions: Dietary Supplement: Green tea
- Fermented green tea (Experimental): Fermented green tea extract 2 gram per day
  Interventions: Dietary Supplement: Green tea
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Green tea

INTERVENTIONS:
Dietary Supplement: Green tea — We made a dietary supplement from Cammellia sinesis O. Kunze, and made tablets containing extract.

SUMMARY:
The investigators randomly assigned green tea extract, fermented green tea extract, or placebo in adult subjects whose BMI was 25-35 kg/m2. Participants were 40 in each group, and treatment duration was 12 weeks. Primary outcomes were body weight change and fat mass change from baseline to 12 weeks, and secondary outcomes were metabolic parameteres and gut microbiota.

DETAILED DESCRIPTION:
After screening obese subjects who met the inclusion and exclusion criteria, the investigators randomly assigned the two treatment arms and one placebo arm at 1:1:1 ratio. At baseline, anthropometric and biochemical evaluations were conducted including body weight, body composition (DXA and Fat CT), lipid profiles, and liver function test. The tablets were supplied to each participants under double-blind conditions. The investigators obtained blood and stool samples both baseline and final visit at 12 weeks. For improving compliance for treatments, the investigators checked diary for lifestyle and drug compliance every 6 week.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60 years
* BMI 25-35 kg/m2
* Abdominal obesity (Waist circumference): Male >90 cm, Female >85cm

Exclusion Criteria:

* Cardiovascular events within 3 months
* uncontrolled hypertension (>160/100 mmHg)
* Diabetes mellitus
* Dyslipidemia under statin therapy
* TSH<0.1 uU/ml or>10 uU/ml
* Elevated creatinine level (twice higher than upper normal limit)
* Elevated AST/ALT level (three times higher than upper normal limit)
* Pregnancy, lactation

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03-20 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Body weight | Baseline, and 12 weeks
  Body weight change were calculated using electronic scale
Body fat | Baseline, and 12 weeks
  Total body fat change were calculated using DXA and abdominal fat CT

SECONDARY OUTCOMES:
Waist circumference | Baseline, 6 weeks, and 12 weeks
  Waist circumference was measured using standard method
Lipid profile | Baseline, and 12 weeks
  total cholesterol, TG, HDL-C, LDL-C, TG/HDL-C, Apo B/ApoA1, Apo B, Apo A1
Inflammatory markers | Baseline, and 12 weeks
  hs-CRP, ESR, inflammatory cytokines (TNFa, IL-1β, IL-6)
Microbiota | Baseline, and 12 weeks
  Gut Microbiota composition